CLINICAL TRIAL: NCT04808804
Title: Retinal Neurodegeneration In Patients With Type 2 Diabetes Mellitus Without Diabetic Retinopathy or With Mild Non Proliferative Diabetic Retinopathy Detected by Optical Coherence Tomography
Brief Title: Retinal Neurodegeneration In Type 2 Diabetes Mellitus Detected by Optical Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emel Saad Tawadrous, Principal Investigator, Assiut University
Other Study IDs: Neurodegeneration In DM
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Retinal Neuropathy; Neurodegeneration
MeSH Terms: conditions — Nerve Degeneration | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DM: Patients With Type 2 Diabetes Mellitus without any signs of diabetic retinopathy or with mild non proliferative diabetic retinopathy
  Interventions: Diagnostic Test: Optical Coherence Tomography (OCT)
- Healthy: healthy controls
  Interventions: Diagnostic Test: Optical Coherence Tomography (OCT)

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography (OCT) — a noninvasive imaging technology used to obtain high resolution cross-sectional images of the retina

SUMMARY:
Evaluation of retinal neurodegeneration in patients with type 2 diabetes mellitus (DM2) without diabetic retinopathy or with mild non proliferative diabetic retinopathy

DETAILED DESCRIPTION:
Retinal complications in diabetes mellitus (DM) patients were typically considered part of a vascular process. However, recent studies suggest that ocular degeneration in DM might be caused by 2 different conditions: vasculopathy and neuropathy . For some authors, neuropathy observed in the retina of DM patients might be a part of an underlying polyneuropathy ; for others, however, neuropathic changes might precede microvascular alterations .

Axons of retinal ganglion cells compose the retinal nerve fiber layer (RNFL) in the retina and then form the optic nerve connecting the eyeball and brain. Retinal nerve fiber layer (RNFL) loss is recognized as an important neurodegenerative sign in glaucoma. Thinning of the RNFL has also been found in multiple sclerosis, Parkinson's disease and Alzheimer's disease, indicating neurodegeneration of the retina. If RNFL thinning is significant in diabetic patients with preclinical diabetic retinopathy, evaluation of peripapillary RNFL thickness would be very important, because early detection and treatment of diabetic retinopathy is critical to reduce the risk of blindness Optical coherence tomography (OCT) has been introduced into clinical practice as the most noninvasive and objective method to visualize the retina, showing an amount of detail that resembles histological specimens. Initially, OCT was applied to detect complications of DR (edema macular or epiretinal membrane). Later on, it allowed quantitative and qualitative measurements of retinal thickness and segmentation of all intraretinal layers. OCT might detect early retinal neurodegenerative changes, and thus help define which diabetic patients may be at risk to develop DR.

ELIGIBILITY:
Inclusion Criteria:

* All patients with confirmed type 2 DM diagnosis of at least 6 months
* Best-corrected visual acuity (BCVA) of 6/12 or higher (using a Snellen chart) in each eye
* Intraocular pressure (by applanation) less than 21 mmHg.
* Healthy controls had no record nor evidence of ocular or neurologic disease of any kind; their BCVA is > 6/9 based on the Snellen scale.

Exclusion Criteria:

* presence or past history of moderate or severe non proliferative diabetic retinopathy or proliferative diabetic retinopathy , confirmed by indirect funduscopy or retinography images.
* presence of significant refractive errors (≥5 diopters of spherical equivalent refraction or 3 diopters of astigmatism)
* intraocular pressure ≥21 mmHg
* media opacifications
* concomitant ocular diseases, including history of glaucoma or retinal pathology
* systemic conditions that could affect the visual system, including neurodegenerative disorders such as Parkinson's disease, multiple sclerosis, or dementia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 eyes of patients with DM2 and without any signs of diabetic retinopathy or with mild non proliferative diabetic retinopathy and 40 eyes of healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
RNFL thickness | Baseline
  retinal nerve fiber layer (RNFL) will be evaluated

REFERENCES:
- [Background] Santos AR, Ribeiro L, Bandello F, Lattanzio R, Egan C, Frydkjaer-Olsen U, Garcia-Arumi J, Gibson J, Grauslund J, Harding SP, Lang GE, Massin P, Midena E, Scanlon P, Aldington SJ, Simao S, Schwartz C, Ponsati B, Porta M, Costa MA, Hernandez C, Cunha-Vaz J, Simo R; European Consortium for the Early Treatment of Diabetic Retinopathy (EUROCONDOR). Functional and Structural Findings of Neurodegeneration in Early Stages of Diabetic Retinopathy: Cross-sectional Analyses of Baseline Data of the EUROCONDOR Project. Diabetes. 2017 Sep;66(9):2503-2510. doi: 10.2337/db16-1453. Epub 2017 Jun 29. PMID 28663190
- [Background] Shahidi AM, Sampson GP, Pritchard N, Edwards K, Vagenas D, Russell AW, Malik RA, Efron N. Retinal nerve fibre layer thinning associated with diabetic peripheral neuropathy. Diabet Med. 2012 Jul;29(7):e106-11. doi: 10.1111/j.1464-5491.2012.03588.x. PMID 22269030
- [Background] Salvi L, Plateroti P, Balducci S, Bollanti L, Conti FG, Vitale M, Recupero SM, Enrici MM, Fenicia V, Pugliese G. Abnormalities of retinal ganglion cell complex at optical coherence tomography in patients with type 2 diabetes: a sign of diabetic polyneuropathy, not retinopathy. J Diabetes Complications. 2016 Apr;30(3):469-76. doi: 10.1016/j.jdiacomp.2015.12.025. Epub 2015 Dec 30. PMID 26809902
- [Background] Simo R, Hernandez C; European Consortium for the Early Treatment of Diabetic Retinopathy (EUROCONDOR). Neurodegeneration in the diabetic eye: new insights and therapeutic perspectives. Trends Endocrinol Metab. 2014 Jan;25(1):23-33. doi: 10.1016/j.tem.2013.09.005. Epub 2013 Nov 1. PMID 24183659
- [Background] Zangwill LM, Bowd C. Retinal nerve fiber layer analysis in the diagnosis of glaucoma. Curr Opin Ophthalmol. 2006 Apr;17(2):120-31. doi: 10.1097/01.icu.0000193079.55240.18. PMID 16552246
- [Background] Petzold A, de Boer JF, Schippling S, Vermersch P, Kardon R, Green A, Calabresi PA, Polman C. Optical coherence tomography in multiple sclerosis: a systematic review and meta-analysis. Lancet Neurol. 2010 Sep;9(9):921-32. doi: 10.1016/S1474-4422(10)70168-X. PMID 20723847
- [Background] Satue M, Garcia-Martin E, Fuertes I, Otin S, Alarcia R, Herrero R, Bambo MP, Pablo LE, Fernandez FJ. Use of Fourier-domain OCT to detect retinal nerve fiber layer degeneration in Parkinson's disease patients. Eye (Lond). 2013 Apr;27(4):507-14. doi: 10.1038/eye.2013.4. Epub 2013 Feb 22. PMID 23429414
- [Background] Marziani E, Pomati S, Ramolfo P, Cigada M, Giani A, Mariani C, Staurenghi G. Evaluation of retinal nerve fiber layer and ganglion cell layer thickness in Alzheimer's disease using spectral-domain optical coherence tomography. Invest Ophthalmol Vis Sci. 2013 Sep 5;54(9):5953-8. doi: 10.1167/iovs.13-12046. PMID 23920375
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] van Dijk HW, Verbraak FD, Stehouwer M, Kok PH, Garvin MK, Sonka M, DeVries JH, Schlingemann RO, Abramoff MD. Association of visual function and ganglion cell layer thickness in patients with diabetes mellitus type 1 and no or minimal diabetic retinopathy. Vision Res. 2011 Jan 28;51(2):224-8. doi: 10.1016/j.visres.2010.08.024. Epub 2010 Aug 27. PMID 20801146
- [Background] Fischer MD, Huber G, Beck SC, Tanimoto N, Muehlfriedel R, Fahl E, Grimm C, Wenzel A, Reme CE, van de Pavert SA, Wijnholds J, Pacal M, Bremner R, Seeliger MW. Noninvasive, in vivo assessment of mouse retinal structure using optical coherence tomography. PLoS One. 2009 Oct 19;4(10):e7507. doi: 10.1371/journal.pone.0007507. PMID 19838301
- [Background] Ceklic L, Maar N, Neubauer AS. Optical coherence tomography fast versus regular macular thickness mapping in diabetic retinopathy. Ophthalmic Res. 2008;40(5):235-40. doi: 10.1159/000127830. Epub 2008 Apr 25. PMID 18437033
- [Background] Wilkinson CP, Ferris FL 3rd, Klein RE, Lee PP, Agardh CD, Davis M, Dills D, Kampik A, Pararajasegaram R, Verdaguer JT; Global Diabetic Retinopathy Project Group. Proposed international clinical diabetic retinopathy and diabetic macular edema disease severity scales. Ophthalmology. 2003 Sep;110(9):1677-82. doi: 10.1016/S0161-6420(03)00475-5. PMID 13129861